CLINICAL TRIAL: NCT02814630
Title: Three-month, Single-center Study to Identify Biomarkers (Plasma Exosomal miRNAs) and Mechanism of Response (Basophil Transcriptome Analysis) to Xolair® (Omalizumab) in Patients With Chronic Idiopathic Urticaria
Brief Title: Three-month, Single-center Study to Identify Biomarkers/Response to Xolair Therapy in Chronic Idiopathic Urticaria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asthma Inc Clinical Research Center (Other)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIGE025EUS44T
Record Dates: First submitted 2016-05-31; First posted 2016-06-28 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Chronic Idiopathic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label Xolair (Other): The patients will receive one subcutaneous injection of omalizumab at a dose of 300 mg on Days 1, 30, and 60.
  There is no control drug.
  Interventions: Biological: Xolair

INTERVENTIONS:
Biological: Xolair — The patients will receive one subcutaneous injection of Xolair® (omalizumab) at a dose of 300 mg on Days 1, 30, and 60. This dose is based on the results of the international, multicenter, randomized, double-blind, placebo-controlled study which demonstrated that omalizumab significantly decreased clinical symptoms and signs of chronic idiopathic urticaria in patients who had remained symptomatic despite the use of H1-antihistamines (Maurer et al., 2013)
  Other Names: Omalizumab

SUMMARY:
This is a single center, non-comparative exploratory study, to investigate the effect of omalizumab over a 3-month treatment period in adult (≥18 years) patients with chronic idiopathic urticaria who had remained symptomatic despite the use of high dose H1-antihistamines.

DETAILED DESCRIPTION:
This is a single center, non-comparative exploratory study, to investigate the effect of omalizumab over a 3-month treatment period in adult (≥18 years) patients with chronic idiopathic urticaria who had remained symptomatic despite the use of high dose H1-antihistamines. After an initial screening visit within two weeks of the Day 1 baseline visit, patients receive one subcutaneous injection of omalizumab at a dose of 300 mg on Days 1, 30, and 60. Patients will return for clinical assessments and blood draws on Day 3 and Day 30 (study conclusion). Blood will be collected at the screening visit (Day -14), baseline (Day 1, prior to omalizumab injection), Day 14, Day 30 (prior to omalizumab injection), Day 60 (prior to omalizumab injection), and Day 90 (study completion) for microsomal miRNA extraction, basophil isolation, and also stored at -70oC for later periostin assays for a total of 275ml of blood over the course of the study (25ml at screening and 50ml for each of the 5 subsequent visits (i.e., Days 1, 14, 30, 60, and 90). Plasma exosomal miRNA bioinformatics analyses will be conducted in early (i.e., Day 14) and later (i.e., Day 30, 60, 90) responder groups. The 2 wk time point will capture the early responders and the 4, 8, and 12 wk time points will capture the remaining responder groups based on the following: Two Phase III, global, multicenter, randomized, double-blind, placebo-controlled trials (Appendix B, CIU Study 1 and CIU Study 2 data) and data of CIU patients with a starting UAS7 score of 25.3 ± 2.0 (mean ± SEM) treated with Xolair® outside of clinical trials (Metz et al., 2014), where 57% attained complete response within one week of their first treatment and a further 29% within 4 weeks (Metz et al., 2014).

To address the role/mechanism of basophils in the immunopathogenesis of chronic urticaria, we will do basophil mRNA/miRNA arrays.

ELIGIBILITY:
Inclusion Criteria:

* • at least 6 weeks of chronic idiopathic urticaria with itching despite current use of up to x4 H1-antihistamines (Kaplan, 2004)

  * an urticaria activity score (UAS) during a 7-day period (UAS7) of 16 or more (on a scale ranging from 0 to 42, with higher scores indicating greater activity and a minimally important difference [MID] of 9.5 to 10.5) (Mathias et al., 2012)
  * a weekly itch-severity score (ISS) of 8 or more (on a scale ranging from 0 to 21, with higher scores indicating more severe itching and an MID of ≥5) during the 7 days before first treatment with omalizumab.
  * All females of childbearing potential must be either abstinent from sexual intercourse or using adequate contraception and must also have a negative urine pregnancy test.*

Exclusion Criteria:

* • a clearly defined underlying cause for chronic urticaria (e.g., physical urticaria)

  * routine administration (i.e., daily or every other day for ≥5 consecutive days) of systemic glucocorticoids, hydroxychloroquine, methotrexate, cyclosporine, cyclophosphamide, or intravenous immune globulin within the previous 30 days
  * the use of any H2-antihistamine or leukotriene-receptor antagonist within 7 days preceding the screening visit
  * a history of cancer
  * a known hypersensitivity to omalizumab
  * treatment with omalizumab within the previous year, or
  * pregnant or nursing females*

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

PRIMARY OUTCOMES:
miRNAs in the blood differentially expressed after treatment with Xolair® in patients with chronic idiopathic urticaria. | 12 week period of Xolair® treatment
  Identification of specific miRNA(s) that are novel biomarker(s) predicting response to Xolair® treatment in 20 patients with chronic idiopathic urticaria.

CONTACTS AND LOCATIONS:
Overall Officials: William Henderson, MD, Study Director — University of Washington
Locations (1):
- ASTHMA Inc Clinical Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
A paper may be written but individual participant data will not be made available